CLINICAL TRIAL: NCT05239650
Title: An Open-label, Multicenter, Phase II Clinical Study to Evaluate the Efficacy and Safety of HLX07 (Recombinant Humanized Anti-EGFR Monoclonal Antibody Injection) + HLX10 (Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection) + mFOLFOX6 or HLX07 Monotherapy in Patients With Metastatic Colorectal Cancer
Brief Title: Phase II Clinical Study to Evaluate the Efficacy and Safety of HLX07+HLX10 +mFOLFOX6 or HLX07 Monotherapy in Patients With mCRC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX07-mCRC201
Record Dates: First submitted 2022-02-07; First posted 2022-02-15 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-02

CONDITIONS: CRC
MeSH Terms: interventions — HLX07

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A：1L treatment (Experimental): HLX07 * 1000 mg+HLX10* 200mg +mFOLFOX6, IV, Q2W
  Interventions: Drug: HLX07; Drug: HLX10; Drug: mFOLFOX6
- B：≥2L treatment (Experimental): HLX07 *1000 mg monotherapy,IV, Q2W
  Interventions: Drug: HLX07

INTERVENTIONS:
Drug: HLX07 — 1000mg
Drug: HLX10 — 200mg
  Arms: A：1L treatment
Drug: mFOLFOX6 — OXA：85 mg/m2;LV:400 mg/m2；5-FU：400 mg/m2
  Arms: A：1L treatment

SUMMARY:
This is An Open-label, Multicenter, Phase II Clinical Study to Evaluate the Efficacy and Safety of HLX07 (Recombinant Humanized Anti-EGFR Monoclonal Antibody Injection) + HLX10 (Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection) + mFOLFOX6 or HLX07 Monotherapy in Patients with Metastatic Colorectal Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age>=18Y and ≤75Y
* Good Organ Function
* Expected survival time ≥ 3 months
* mCRC that have been diagnosed histologically
* KRAS/NRAS/BRAF WT verified by PCR or NGS of tumor tissue
* ECOG score 0-1;

Exclusion Criteria:

* HIV infection
* Active clinical severe infection;
* A history of other malignancies within two years, except for cured carcinoma in situ of the cervix or basal cell carcinoma of the skin.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 3 years
  Objective response rate (assessed by investigator per RECIST V1.1)
PFS | : from the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier)，up to 3 years
  Progression-free survival (PFS) (assessed by the investigator per RECIST v1.1 )

SECONDARY OUTCOMES:
OS | up to 5 years
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Peng Junjie, Principal Investigator — Fudan University Affiliated Oncology Hospital

IPD SHARING:
Plan to Share IPD: No